CLINICAL TRIAL: NCT05283473
Title: Serum Concentration of Magnesium Attained in Magnesium Sulfate Therapy in Pregnant Women With Severe Preeclampsia
Brief Title: Serum Magnesium Concentration in Magnesium Sulfate Therapy for Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 01/22/DD-BVMD
Record Dates: First submitted 2022-02-12; First posted 2022-03-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-03

CONDITIONS: Severe Pre-Eclampsia
Keywords: Pre-eclampsia; Magnesium sulfate; Eclampsia; magnesium concentration
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pregnant women diagnosed with pre-eclampsia with severe features will be treated with magnesium sulfate to prevent seizures. Magnesium sulfate will be administered according to My Duc Hospital's protocol for treatment of pre-eclampsia (a loading dose of 4.5g given intravenously in 20 min, followed by a maintenance dose at an infusion rate of 1.5g/h). Serum magnesium concentrations will be measured before the loading dose and 0.5h, 1h, 2h, and every 6 hours thereafter.

DETAILED DESCRIPTION:
This observational, longitudinal, prospective case-series aims to assess serum magnesium concentrations at specific times in pregnant women treated with magnesium sulfate for pre-eclampsia with severe features.

Pregnant women aged minimum 18 who are admitted to My Duc Hospital with severe pre-eclampsia, as defined by the American College of Obstetricians and Gynecologists (ACOG) diagnosis criteria, will be indicated for therapy with magnesium sulfate. Only those who give written informed consent will be included in the study. According to the ACOG criteria, pre-eclampsia is considered severe if present with any of the following features : systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110 mmHg, thrombocytopenia (<100,000/mm3) abnormal liver function (increase in transaminases to twice the normal value or pain in the upper right quadrant/epigastrium that is unresponsive to medication), abnormal renal function (creatinine >1.1 mg/dl or twice normal values), acute pulmonary edema and/or new cerebral and/or visual symptoms.

Exclusion criteria includes impaired renal function (eGFR < 60 mL/min/ 1,73 m2 or oliguria ), known hypersensitivity to the drug, severe myasthenia, atrioventricular block or a diminished level of consciousness.

All patients will be given the standard loading dose of 4.5 grams of magnesium sulfate administered over 20 minutes, followed by a maintenance dose of magnesium sulfate at an infusion rate of 1.5g/h, in compliance with My Duc Hospital's guidelines. Maternal blood samples will be obtained for serum magnesium and creatinine concentrations at baseline prior to magnesium sulfate administration; at 30 min, 1 hour, 2 hours, 4 hours and every 6 hours until discontinuation of magnesium sulfate therapy. Antihypertensive medications can be given according to My Duc Hospital's guidelines.

Patients can choose to withdraw from the study at any point without affect on the course of treatment. Investigators can also offer patients to opt out of the study for medical emergencies.

Magnesium sulfate therapy will be discontinued if there is any sign of magnesium toxicity, or the patient has been stable for 24 hours of treatment without any severe hypertensive episode or convulsion.

All patients will be followed up until delivery and both mother and neonate are discharged to record obstetric and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Aged ≥ 18
* Diagnosed with pre-eclampsia with severe features, with or without chronic hypertension, as defined by the American College of Obstetricians and Gynecologists (ACOG) diagnosis criteria.
* Provision of written informed consent to participate as shown by a signature on the patient consent form.

Exclusion Criteria:

* Impaired renal function (eGFR < 60 mL/min/ 1,73 m2 or oliguria )
* Occurrence of eclampsia before magnesium sulfate administration
* Known hypersensitivity to the drug,
* Severe myasthenia, atrioventricular block
* A diminished level of consciousness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged minimum 18 who are admitted to My Duc Hospital with severe pre-eclampsia, as defined by the American College of Obstetricians and Gynecologists (ACOG) diagnosis criteria, and indicated for therapy with magnesium sulfate will be included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Serum magnesium concentrations before and during magnesium sulfate infusion | From administration of loading dose until termination of magnesium sulfate treatment or occurrence of magnesium toxicity, whichever comes first, approximately up to 36 hours.
  Serum magnesium concentrations are measured immediately before the loading dose of magnesium sulfate and at 30 min, 1 hr, 2 hr, 4 hr, 6 hr and then every 6 hours during magnesium sulfate infusion.

SECONDARY OUTCOMES:
Adverse drug reaction | From administration of loading dose until termination of magnesium sulfate treatment or occurrence of magnesium toxicity, whichever comes first, approximately up to 36 hours.
  Rates of adverse drug reactions to administration of magnesium sulfate
Magnesium toxicity | From administration of loading dose until termination of magnesium sulfate treatment or occurrence of magnesium toxicity, whichever comes first, approximately up to 36 hours.
  Rates of patients having signs of magnesium toxicity
Mode of delivery | At birth
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Gestational age at delivery | At birth
  Gestational age at delivery
Rate of preterm birth before 28 weeks of gestation | From date of enrollment until 27 6/7 weeks
  Birth before 28 weeks
Rate of preterm birth before 34 weeks of gestation | From date of enrollment until 33 6/7 weeks
  Birth before 34 weeks
Rate of all live births at any gestational age | At birth
  The birth of at least one newborn, regardless of gestational age, that exhibits any sign of life such as respiration, heartbeat, umbilical pulsation or movement of voluntary muscles
Rate of maternal mortality | From date of enrollment until date of discharge, up to 12 weeks
  Death of the mother
Rate of eclampsia | From date of enrollment until date of discharge, up to 12 weeks
  Onset of seizures (convulsions) in a patient with pre-eclampsia
Rate of HELLP syndrome | From date of enrollment until date of discharge, up to 12 weeks
  The clinical presentation of hemolysis, elevated liver enzymes, and low platelet count in a patient with pre-eclampsia
Rate of placental abruption | From date of enrollment until date of delivery, up to 12 weeks
  Separation of placenta from the inner wall of the uterus before birth
Rate of postpartum hemorrhage | Within 24 hours after delivery
  A cumulative blood loss of greater than or equal to 1,000 mL or blood loss accompanied by signs or symptoms of hypovolemia within 24 hours after the birth process
Rate of stroke | From date of enrollment until date of discharge, up to 12 weeks
  Occurrence of stroke in a patient with pre-eclampsia
Rate of acute kidney injury | From date of enrollment until date of discharge, up to 12 weeks
  A sudden episode of kidney failure or kidney damage that happens within a few hours or a few days in a patient with pre-eclampsia
Rate of liver capsule hematoma or rupture | From date of enrollment until date of discharge, up to 12 weeks
  Occurrence of hepatic rupture or hematoma in a patient with pre-eclampsia
Rate of pulmonary edema | From date of enrollment until date of discharge, up to 12 weeks
  Accumulation of excess fluid in the lungs of a patient with pre-eclampsia
Rate of stillbirth | After 20 weeks of gestation until the date of delivery
  Infant born with no sign of life at or after 20 weeks' gestation
Birthweight | At birth
  Weight of infant born
Rate of small-for-gestational-age | At birth
  Babies born with birthweights below the 10th percentile for babies of the same gestational age.
5-minute Apgar score | At birth
  Apgar score at 5 minute after birth. 5-minute Apgar score of 7-10 as reassuring, a score of 4-5 as moderately abnormal, and a score of 0-3 as low in the term infant and late-preterm infant.
Rate of admission to the neonatal intensive care unit (NICU) | Up to 28 days of life after the due date
  Admission of infant to the neonatal intensive care unit
Rate of death before discharge | Up to 28 days of life after the due date
  Death of newborn before discharge from nursery
Rate of respiratory distress syndrome | Up to 28 days of life after the due date
  Presence of tachypnoea, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Rate of proven sepsis | Up to 28 days of life after the due date
  The combination of clinical signs and positive blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam